CLINICAL TRIAL: NCT07212920
Title: Physiotherapeutic Function-Based Assessment and Diagnosis of Subacute Knee Injuries During Physical or Video-Based Consultations - A Validity and Reliability Study
Brief Title: Validity and Reliability of Video-Based Functional Physiotherapy Assessment of Subacute Knee Injuries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PTassessment_digital_knee
Record Dates: First submitted 2025-08-18; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-08

CONDITIONS: Knee Pain
Keywords: Physiotherapy; Physical therapy; Assessment; Diagnosis; Digital care; Telemedicine; Knee pain; Anterior cruciate ligament; Knee osteoarthritis; Meniscus tears; Collateral ligament
MeSH Terms: conditions — Disease; Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digital assessment first, then face-to-face (Experimental): Participants undergo two knee assessments: one video-based and one in-person. The video-based exam includes standardized history taking and functional tests without specific knee tests, conducted via clinic software with the physiotherapist in a separate room. The in-person exam follows immediately and includes the same functional tests plus specific knee tests (e.g., ligament, meniscus). After each part, physiotherapists assess whether sufficient information is available to proceed with treatment. All assessments follow standardized protocols, pilot-tested by physiotherapists. Data collection occurs at a public rehab clinic in Västra Götaland, with physiotherapists trained prior to study start.
  Interventions: Diagnostic Test: Physiotherapy digital assessment; Diagnostic Test: Physiotherapy assessment - only functional tests

INTERVENTIONS:
Diagnostic Test: Physiotherapy digital assessment — This study involves three types of knee assessments to evaluate diagnostic reliability and validity: (1) a video-based function-based examination without specific knee tests, (2) traditional in-person function-based examination without specific knee tests and to control with (3) a traditional in-person examination including specific knee tests. The video-based assessment includes standardized history taking and functional evaluation conducted via clinic software, with the physiotherapist and participant in separate rooms. Physiotherapists provide diagnostic judgments after each assessment phase. All procedures follow standardized protocols, pilot-tested and conducted at a public rehabilitation clinic in Västra Götaland.
Diagnostic Test: Physiotherapy assessment - only functional tests — This study involves three types of knee assessments to evaluate diagnostic reliability and validity: (1) a video-based function-based examination without specific knee tests, (2) traditional in-person function-based examination without specific knee tests and to control with (3) a traditional in-person examination including specific knee tests. The in-person assessments (2 and 3) includes the same functional tests plus specific tests targeting knee structures (ligaments, meniscus etc). Physiotherapists provide diagnostic judgments after each assessment phase. All procedures follow standardized protocols, pilot-tested and conducted at a public rehabilitation clinic in Västra Götaland.

SUMMARY:
This study aims to validate a function-based physiotherapy assessment for subacute knee pain without using specific knee tests. Assessments are conducted either in-person or via video consultations in primary care. The study also compares the reliability of digital versus physical assessments to determine if video-based evaluations can provide sufficient diagnostic support and guide treatment decisions.

The main questions this study aims to answer are:

1. Is a function-based knee assessment without specific knee tests valid compared to traditional in-person diagnostics using specific tests?
2. Is a video-based assessment based on history and function-based knee assessment without specific knee tests as valid and reliable as an in-person function-based knee assessment?
3. What is the interrater agreement of function-based knee assessments conducted via video compared to those conducted in person?

DETAILED DESCRIPTION:
BACKGROUND Knee pain is one of the most common complaints in primary care. Traditional knee assessments include history-taking, evaluation of joint mobility and muscle strength, and specific tests targeting structures such as ligaments and menisci. However, functional tests-such as chair rise or single-leg stance-evaluate the integrated performance of multiple structures and may be more feasible in digital consultations.

Existing literature shows variable validity for specific knee tests, with only a few reaching acceptable thresholds for sensitivity and specificity. In video-based assessments, joint mobility evaluation is reliable, and functional tests are recommended over strength tests. While some knee tests are suggested for digital use, their measurement properties as self-administered tests under physiotherapist supervision remain unclear.

This study will investigate whether a function-based assessment without specific knee tests can provide sufficient diagnostic information and guide treatment decisions for subacute knee injuries. It will also compare the validity and reliability of digital versus in-person physiotherapy assessments in primary care.

METHODS Participants will be consecutively recruited from public and private rehabilitation clinics in the Västra Götaland region of Sweden. Individuals with subacute knee pain (onset between 1 week and 3 months) will be informed about the study through clinics, websites, and online booking systems. Interested individuals will complete a digital screening form to assess eligibility. Those who meet the inclusion criteria will receive written study information and will be able to provide informed consent digitally via Bank-ID.

Demographic data will be collected through the same form, including age, gender, origin, symptom experience, pain intensity and duration, prior video consultation experience, perceived balance, and estimated travel distance to the clinic. This information will support analysis of environmental and accessibility factors.

Eligible participants will be contacted to schedule two knee assessments-one in-person and one via video. Each visit is expected to last approximately 30 minutes, with additional time allocated for preparation and documentation by the physiotherapists.

Inclusion criteria will include age ≥18, subacute knee symptoms, ability to bear weight and flex the knee, no tenderness over patella or fibula, sufficient Swedish language skills, and access to digital technology.

Exclusion criteria will include prior assessment for current symptoms, recent knee or hip surgery, and inability to walk independently.

Sample size calculations indicate that at least 22 participants per diagnostic category (total n=110) will be needed to detect a kappa coefficient of 0.60. With an estimated 20% dropout rate, the target sample size will be 138. Recruitment will continue until minimum group sizes are met or for up to one year.

The study will evaluate the validity and reliability of function-based knee assessments without specific tests, comparing in-person and video-based formats.

Participants will undergo two consecutive knee assessments at a rehabilitation clinic. The first will be a video-based evaluation, including history-taking and functional tests, conducted in real time with the physiotherapist in a separate room. The second will be a traditional in-person assessment, including both functional and specific knee tests. Physiotherapists will use standardized protocols and receive training prior to data collection.

Data collection Participant background data (e.g., age, gender, pain intensity, duration, prior video visit experience, and travel distance) will be collected via a secure web form after consent. Each participant will undergo two knee assessments-first via video, then in person-conducted by the same physiotherapist. Diagnostic agreement between methods will be evaluated, along with physiotherapist confidence and patient satisfaction. Standardized tools include NRS for pain and KOOS-12 for function and quality of life. Secondary outcomes include adverse events, need for further testing or referral, and time required per visit.

Statistical Analysis:

Descriptive statistics will include means, medians, standard deviations, and quartiles. The in-person assessment with specific knee tests will serve as the gold standard. Diagnostic agreement between methods will be analyzed using Cohen's kappa, which will also be used to assess intra-rater agreement. Sensitivity and specificity will be calculated to evaluate the accuracy of assessments without specific tests. Confidence intervals for kappa values will be reported.

Differences in diagnostic certainty level will be analyzed using paired t-test if the data is normally distributed, and wilcoxon signed-rank test if using non-parametric test.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Subacute knee symptoms (onset more than one week ago but less than three months ago)
* Fulfillment of Ottawa Knee Rule criteria to exclude fractures:

A) Able to bear weight for at least four steps both immediately after injury and at the time of assessment (limping allowed) B) Able to flex the knee to 90 degrees C) No tenderness over the fibular head or patella

* Sufficient proficiency in written and spoken Swedish to complete forms and describe symptoms; no need for interpreter
* Access to digital technology (e.g., computer or smartphone)

Exclusion Criteria:

* Prior assessment for current knee symptoms (by rehab clinic, physician, emergency care, or urgent care)
* Knee or hip replacement surgery within the past year
* Other knee surgeries (ACL, meniscus, ligament) within the past year
* Inability to walk independently, with or without walking aids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Agreement in Diagnostic Categories from Functional In-Person Assessment | Day 1
  Primary outcome is whether the system-level diagnosis (diagnostic category) assigned by the physiotherapist matches across in-person assessments with or without specific tests - functional assessment compared to traditional assessment with specific tests. Diagnoses are categorized into five predefined groups: ligament, meniscus, joint-related, soft tissue, and other. Within each category, physiotherapists assign specific ICD-10 codes. Outcome is measured as match/mismatch between diagnostic categories.
Number of Participants with Agreement in Diagnostic Categories - Digital Assessment Based on Patient History | Day 1
  Primary outcome is whether the system-level diagnosis (diagnostic category) assigned by the physiotherapist matches across digital assessment with only patient history compared with traditional in person assessment with specific tests. Diagnoses are categorized into five predefined groups: ligament, meniscus, joint-related, soft tissue, and other. Within each category, physiotherapists assign specific ICD-10 codes. Outcome is measured as match/mismatch between diagnostic categories.
Number of Participants with Agreement in Diagnostic Categories - Digital Assessment Based on Patient History and Functional Evaluation | Day 1
  Primary outcome is whether the system-level diagnosis (diagnostic category) assigned by the physiotherapist matches across digital assessment with traditional in person assessment with specific tests. Diagnoses are categorized into five predefined groups: ligament, meniscus, joint-related, soft tissue, and other. Within each category, physiotherapists assign specific ICD-10 codes. Outcome is measured as match/mismatch between diagnostic categories.
Number of participants with agreement in test results of functional assessment | Day 1
  Primary outcome is whether the test results from the functional tests performed in the video consultation differs from in-person functional assessment.

SECONDARY OUTCOMES:
Degree of diagnostic certainty | Day 1
  After each assessment, the physiotherapists will rate their level of diagnostic certainty on a scale from 0 (not confident) to 100 (fully confident), for a total of four ratings.
  A) digital patient history assessment B) digital functional assessment C) in-person functional assessment D) in-person specific tests
Number of Participants with Agreement on Specific Diagnostic Categories | Day 1
  The physiotherapists will diagnose with pre-defined ICD-10 diagnoses. All assessments will be compared on a specific diagnostic level.
Patient-Rated Satisfaction With the Assessment | Day 1
  Patient satisfaction will be measured after each knee assessment session using a modified item from the Swedish instrument "Quality from the Patient's Perspective" (QPP). The selected item is: "I received the best possible examination (as far as I can judge myself)." Patients rate their agreement on a 5-point Likert scale: Strongly agree, Mostly agree, Partly agree, Do not agree at all, and Not applicable. The response is collected via a secure web-based form.
Adverse events | Day 1
Number of Participants Requiring Additional Specific Knee Tests Following Assessment | Day 1
Number of Participants Requiring Supplementary In-Person Examinations After Video-Based Assessment | Day 1
Number of Participants Referred to a Physician Following Assessment | Day 1
Time required for each visit | Day 1
Reliability of 30 seconds chair stand test | Day 1
  The reliability of testing physical function will be evaluated by the physiotherapist during each assessment session, video-based assessment compared with in-person assessment. Participants perform as many sit-to-stand repetitions as possible within 30 seconds, with arms crossed over the chest. One trial repetition is allowed before the test begins. If unable to perform without assistance, hand support may be used. Each repetition must result in a fully upright standing position, with feet remaining on the floor throughout. The total number of correctly performed repetitions is recorded.
Reliability of Joint Mobility Assessment | Day 1
  The reliability of testing joint mobility will be evaluated by the physiotherapist during each assessment session, video-based assessment compared with in-person assessment.The range of motion is rated using a standardized scale with the following categories:
  Impaired Slightly impaired Normal Unable to perform Not assessed
Reliability of Sit-to-Stand Ability From Chair | Day 1
  The reliability of the functional test stand up from sitting will be evaluated by the physiotherapist during each assessment session, video-based compared with in-person assessment. The participant's ability to rise from a chair is assessed using a standardized rating scale:
  Impaired Slightly impaired Normal Unable to perform Not assessed
  Assessment is based on movement quality, control, and ability to complete the task without assistance. The rating is performed by a physiotherapist during each session.
Reliability of Lunge Performance | Day 1
  The reliability of testing functional performance through forward lunge will be evaluated by the physiotherapist during each assessment session, video-based assessment compared with in-person assessment. The participant's ability to perform a forward lunge is assessed using a standardized rating scale:
  Impaired Slightly impaired Normal Unable to perform Not assessed
  Assessment is based on movement control, balance, depth, and ability to complete the task without assistance. The rating is performed by a physiotherapist during each session.
Reliability of Single-Leg Squat Performance | Day 1
  The reliability of testing physical performance through single-leg squat will be evaluated by the physiotherapist during each assessment session, video-based assessment compared with in-person assessment. The participant's ability to perform a single-leg squat is assessed using a standardized rating scale:
  Impaired Slightly impaired Normal Unable to perform Not assessed
  Assessment focuses on movement control, knee alignment, depth, and ability to complete the task without assistance. The rating is performed by a physiotherapist during each session.
Reliability of Sit-to-Stand Ability From Chair | Day 1
  The reliability of testing physical performance through standing up from sitting on a chair will be evaluated by the physiotherapist during each assessment session, video-based assessment compared with in-person assessment. The participant's ability to rise from a chair is assessed using a standardized rating scale:
  Impaired Slightly impaired Normal Unable to perform Not assessed
  Assessment is based on movement quality, control, and ability to complete the task without assistance. The rating is performed by a physiotherapist during each session.
Reliability of Heel Raise Performance | Day 1
  The reliability of testing physical performance through heel raises will be evaluated by the physiotherapist during each assessment session, video-based assessment compared with in-person assessment. The participant's ability to perform heel raises is assessed using a standardized rating scale:
  Impaired Slightly impaired Normal Unable to perform Not assessed
  Assessment is based on movement control, range, and ability to complete the task without assistance. The rating is performed by a physiotherapist during each session.

OTHER OUTCOMES:
Demographic data | At baseline before physiotherapy assessment
  Background information about each participant will be collected. Collected data includes age, sex, origin, height, weight, experience of knee symptoms, pain intensity, pain duration, previous experience with video consultations, travel distance (in kilometers) between home/start point and the clinic, and results from the knee assessments. Travel distance is recorded to enable analysis of transport and environmental aspects.
Knee Pain Intensity Measured by Numeric Rating Scale (NRS) | At baseline before physiotherapy assessment
  Pain intensity will be assessed using the Numeric Rating Scale (NRS), where participants rate their current knee pain, average pain over the past week, and the lowest and highest pain intensity experienced during the past week. Ratings are given on a scale from 0 (no pain) to 10 (worst imaginable pain). NRS has strong correlation with the Visual Analog Scale (VAS) and demonstrates high reliability (intraclass correlation coefficient = 0.95). The minimal detectable change is 1.3.
Knee Injury and Osteoarthritis Outcome Score - 12 Items (KOOS-12) | At baseline before physiotherapy assessment
  KOOS-12 is a shortened version of the original KOOS instrument, consisting of 12 items across three dimensions: pain, function, and quality of life. Each item is scored from 0 (no problems) to 4 (extreme problems). Scores for each dimension are summed and converted to a 0-100 scale, where lower scores indicate more severe symptoms and higher scores indicate milder symptoms. KOOS-12 has demonstrated good reliability, validity, and responsiveness.

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will not be publicly shared due to restrictions under the EU General Data Protection Regulation (GDPR). However, anonymized data may be made available upon reasonable request, provided the request complies with GDPR and Swedish data protection regulations. The following study documents will be shared publicly on a Swedish platform R&D Project Database in Region Västra Götaland and can be translated if requested: Study Protocol, Statistical Analysis Plan (SAP), and Informed Consent Form (ICF).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Start: After ethical approval. Anticipated date: October 1st. End: Available as long as R&D Project Database in Region Västra Götaland is available.
Access Criteria: Individual participant data (IPD) will be provided if the request complies with GDPR and Swedish data protection regulations. The following study documents will be shared publicly on a Swedish platform R&D Project Database in Region Västra Götaland and can be translated if requested: Study Protocol, Statistical Analysis Plan (SAP), and Informed Consent Form (ICF).
URL: https://www.researchweb.org/is/se/vgr/project/284257